CLINICAL TRIAL: NCT05658978
Title: Effects of Neuromuscular Training on Selected Physical Fitness Components, Functional Movement, and Handball Skills Among Elite Male Handball Players in Pakistan
Brief Title: Neuromuscular Training on Handball Players Selected Physical Fitness Components, Functional Movement and Handball Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Saddam Akbar, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: GS61103
Record Dates: First submitted 2022-11-19; First posted 2022-12-21 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Inactivity, Physical
Keywords: Physical Fitness Components; Handball Skills; Functional movement; Male Handball Players
MeSH Terms: conditions — Sedentary Behavior | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: In this experiment, the experimental group will continue neuromuscular training exercises and the control group will continue previous regular exercises with coaches' guidelines. Each group has equally male players.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular training of male handball players (Experimental): Neuromuscular training exercises focus on improving physical fitness and skills performance. Neuromuscular training targets the neuromuscular system through engagements of muscle groups as well as nerve function to optimize movements. This training has been considered an effective treatment method to enhance the neurophysiological entity of the joints for coordinated functioning. However, the present study applied neuromuscular training to elite male handball players to assess fitness level as well as skill performance. Post-test 1 will be after 6 weeks, and post-test 2 after 12 weeks to measure performance.
  Interventions: Other: Neuromuscular training
- Male handball players continue previous regular exercises (Active Comparator): Handball players as a control group will be continuing their previous regular exercises for 12 weeks.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Neuromuscular training — Neuromuscular training Length: 12 weeks; Training duration: 90 minutes; Intensity: 70-95%; 3 days per week. The intensity of the training is increasing in the first 20 minutes, and the intensity is gradually decreasing in the next 5 minutes; Rest: 30 seconds rest between exercises and 1-minute rest between sets.
  Arms: Neuromuscular training of male handball players
Other: Control group — The Control group continues previous regular exercises for 12 weeks with a duration of 90 minutes and three days per week.
  Arms: Male handball players continue previous regular exercises

SUMMARY:
The neuromuscular training improves nerve-muscle control while increasing the stability of functioning joints. Furthermore, Neuromuscular training has been proven to influence the sensitivity and reactivity of the central nervous system and improves the power of athletes by targeting motor units and coordinating motor units and increasing muscle activation. These enhancements resulted in skillful movements and significantly improved agility, balance, muscular strength and muscular power among individuals. The neuromuscular training also focuses on promoting functional joint stability by improving athletes' neuromuscular control and has been proven to significantly enhance athletes' performance. Finally, to evaluate that neuromuscular training can improve elite male handball players' physical fitness components, handball skills and functional movement.

DETAILED DESCRIPTION:
This study included two groups, namely the control and neuromuscular training groups. The sample is 18-22-year-old Pakistani elite male handball players who do not do neuromuscular training exercises. Based on the literature review, the training frequency of this experiment was arranged three (3) times/week, the total training duration will be 12 weeks, and the time of each training session will be changed over two weeks. The 12 weeks of exercise last 90 minutes, with a 10-minute warm-up and a 10-minute cool-down. Training intensity ranges from 70% to 95%. Teach all sports techniques before the intervention. In contrast, the control group discussed with their coaches and will continue the 12-week of previous regular exercises.

Content of Experimental Group: Week 1-2: Introduces the classification of neuromuscular training starting from the: One-leg balance and hamstrings and hip flexor each side exercises; Week 3-4: exercises to improve physical fitness: Agility drills ladder hurdles cones, barrier jump forward-backward and Seated press-ups exercises; 5-6 Week: Reviewed the basic handball skills: Net zigzag, baseline-net-baseline (9 cones), balance board stands on one foot to catch the ball (handball) and biceps and triceps, free weights exercises; 7-8 Week: learn the exercises: Mini-arm circles, tennis ball against wall, Swiss ball side plank (Bodyweight) and Iliotibial band each side exercises; 9-10 Week: Review the Sprints: Baseline-net, gastrocnemius/soleus each side, 4-square, various patterns and vertical jump with an additional load exercises; 11-12 Week: Review physical fitness, handball skills and functional movement: Court suicide sprint conditioning drills, Single-leg squats on half foam roll, Push-up with and without countermovement, Plank 3 levels of difficulty, Ladder: various patterns, biceps each side and Single-leg balance with ball handling drills on half foam roll exercises.

ELIGIBILITY:
Inclusion Criteria:

* The population must be elite male handball players between the ages of 18 to 22
* Able to perform all tests and be Physically active (no previous experience performing neuromuscular training)
* Only players who understand the study purposes and procedures and can complete this training requirement can be included in the research data.

Exclusion Criteria:

* Female handball players should be excluded from this study
* On medication that may affect body composition and muscles activity
* Presently engaged in regular neuromuscular training programs
* Players who are consistently late or absent from training sessions will eventually be excluded

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Speed performance of handball players | 2 weeks
  Speed will be measured by a 30-meter sprint test. To monitor the development of the athlete's maximum sprint speed, the 20m sprint test measurement also has a high reliability value (r=0.94 to 0.98).
Agility performance of handball players | 3 weeks
  Agility will be measured by Illinois agility test running agility using various turns and movements. Participants should lie on their front (head to the start line) and hands by their shoulders. On the 'Go' command the stopwatch is started, and the athlete gets up as quickly as possible and runs forwards 10 meters to run around a cone, then back 10 meters, then runs up and back through a slalom course of four cones. Finally, the athlete runs another 10 meters up and back past the finishing cone.
Balance performance of handball players | 4 weeks
  Balance will be measured by the Star excursion balance test (SEBT). Balance ability of athletes on an activity to keep their balance equilibrium. It is a type of dynamic stability testing. The SEBT involves having a participant maintain a base of support with one leg while maximally reaching in different directions with the opposite leg without compromising base of support of stance leg.
Explosive power of handball players | 5 weeks
  To measure the explosive power of the leg in vertical jump height jumped. The player chalks the end of his fingertips, stands side onto the wall, keeping both feet remaining on the ground, reaches up as high as possible with one hand and marks the wall with the tips of the fingers. From a static position jump as high as possible and marks the wall with the chalk on his fingertips.
Flexibility of handball players | 6 weeks
  The test will be conducted indoors using a static sit and reach box, supplied with a tape measure. The participant will give the instruction to sit with legs together and extended in front of him, so that the feet (shoes off) touch the first step. Both knees will be held together and flat on the floor. The purpose of this test is to assess the flexibility of the lower back and hamstring. The intra-class correlation coefficient for test-retest reliability for the sit and reach test was 0.93.
Muscular Strength of handball players | 8 weeks
  Muscular strength will be measured by the 1RM test. Test-retest ICCs ranged from 0.64 to 0.99 (median ICC = 0.97), where 92% of ICCs were ≥ 0.90, and 97% of ICCs were ≥ 0.80. Based on the previous studies, it can be concluded that the 1RM test generally has good to excellent test-retest reliability, part of the body assessed (upper vs. lower body).
Functional Movement of handball players | 9 weeks
  The FMS will be used to assess the study participants using the standard 0-3 ordinal scale. A score of 3 will be awarded for performing the specific movement perfectly, a score of 2 for completing the movement with some compensatory movements observed, a score of 1 for the subject failing to complete the movement, and a score of 0 for the movement being painful. Functional movement assesses through the FMS Kit.
Dribbling skill performance of handball players | 11 weeks
  Slalom sprint and dribble test will measure dribbling performance. Twelve cones will be placed in a zigzag pattern, and the participant is to slalom the 30-m course as fast as possible. Sprints will be timed using a stopwatch. Slalom sprint and dribble test the indication of a good reliability (without ball: Intraclass Correlation Coefficient [ICC] = 0.91; with ball: ICC = 0.79) and validity (i.e., discriminative between level of performances).
Shooting skill performance of handball players | 12 weeks
  Shooting skill performance will be measure by shooting accuracy test. To measure the shooting ability of accuracy for team handball players can make throws at the target in team handball. Each player had eight shots executed from five different positions, previously established, in the direction of the goal.

CONTACTS AND LOCATIONS:
Overall Officials: Saddam Akbar, PhD, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- University of Agriculture, Hub of Handball in Pakistan, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate.

REFERENCES:
- [Background] Barber-Westin SD, Hermeto AA, Noyes FR. A six-week neuromuscular training program for competitive junior tennis players. J Strength Cond Res. 2010 Sep;24(9):2372-82. doi: 10.1519/JSC.0b013e3181e8a47f. PMID 20703159
- [Background] Barber-Westin, S., Hermeto, A., and Noyes, M.D.F. (2015). A six-week neuromuscular and performance training program improves speed, agility, dynamic balance, and core endurance in junior tennis players. J Athl Enhancement 4.
- [Background] Borghuis, A. J., Lemmink, K. A., Hof, A. L., & Visscher, C. 5. The Effect of a Soccer-Specific Neuromuscular Training Program on Stability, Agility and Injury in Elite Youth Soccer. Core Stability in Soccer: it's a Matter of Control! 83.
- [Background] McLeod TC, Armstrong T, Miller M, Sauers JL. Balance improvements in female high school basketball players after a 6-week neuromuscular-training program. J Sport Rehabil. 2009 Nov;18(4):465-81. doi: 10.1123/jsr.18.4.465. PMID 20108849
- [Background] Trajkovic N, Bogataj S. Effects of Neuromuscular Training on Motor Competence and Physical Performance in Young Female Volleyball Players. Int J Environ Res Public Health. 2020 Mar 8;17(5):1755. doi: 10.3390/ijerph17051755. PMID 32182680